CLINICAL TRIAL: NCT05773144
Title: Adaptive Randomization of Aerobic Exercise During Chemotherapy in Colon Cancer
Acronym: ACTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth Translational Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Justin Brown, Senior Investigator, AdventHealth Translational Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PBRC 2022-018; U01CA271279 (NIH)
Record Dates: First submitted 2023-03-06; First posted 2023-03-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Colonic Neoplasms
MeSH Terms: conditions — Colonic Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Attention control (Sham Comparator): Static stretching
  Interventions: Behavioral: Progressive stretching
- 75 min/wk aerobic exercise (Experimental): Aerobic exercise at a dose of 75 minutes per week
  Interventions: Behavioral: Aerobic exercise
- 150 min/wk aerobic exercise (Experimental): Aerobic exercise at a dose of 150 minutes per week
  Interventions: Behavioral: Aerobic exercise
- 225 min/wk aerobic exercise (Experimental): Aerobic exercise at a dose of 225 minutes per week
  Interventions: Behavioral: Aerobic exercise
- 300 min/wk aerobic exercise (Experimental): Aerobic exercise at a dose of 300 minutes per week
  Interventions: Behavioral: Aerobic exercise

INTERVENTIONS:
Behavioral: Aerobic exercise — Moderate- to vigorous-intensity aerobic exercise
  Arms: 150 min/wk aerobic exercise; 225 min/wk aerobic exercise; 300 min/wk aerobic exercise; 75 min/wk aerobic exercise
Behavioral: Progressive stretching — Static stretching of eight major muscle groups
  Arms: Attention control

SUMMARY:
To goal of this clinical trial is to quantify the dose-response effects of aerobic exercise training compared to attention control on chemotherapy relative dose intensity in colon cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically confirmed stage II or III colon cancer
* Completed surgical resection with curative intent
* Plan to initiate chemotherapy
* Engage in <60 minutes per week of moderate- to vigorous-intensity structured aerobic exercise
* No planned major surgery during the study period
* Readiness to exercise, as determined by a modified version of the Physical Activity Readiness Questionnaire
* Can walk 400 meters
* Can read and speak English
* Ability to provide written informed consent
* Provide written approval by qualified healthcare professional
* Willing to be randomized

Exclusion Criteria:

* Evidence of metastatic colon cancer
* Concurrently actively treated other (non-colon) cancer
* Currently pregnant, breastfeeding, or planning to become pregnant within the next 24 weeks
* Currently participating in another study with competing outcomes
* Any other condition that, in the opinion of the investigator, would preclude participation or successful compliance with the protocol
* Any other situation that, in the opinion of the investigator, would negatively impact subject safety or successful compliance with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Chemotherapy Relative Dose Intensity | 12- or 24-weeks
  The ratio of the delivered dose intensity to the standard or planned dose intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Justin C. Brown, Ph.D., Principal Investigator — AdventHealth; Jeffrey A. Meyerhardt, M.D., M.P.H., Principal Investigator — Dana-Farber Cancer Institute; Bette J. Caan, Dr.P.H., Principal Investigator — Kaiser Permanente
Locations (3):
- United States (3):
  - Kaiser Permanente Northern California, Oakland, California
  - AdventHealth, Orlando, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes